CLINICAL TRIAL: NCT03790553
Title: A Phase III Study of Comparing 61.2 Gy Radiotherapy Dose Versus 50.4 Gy Radiotherapy Dose for Locally Advanced Esophageal Carcinoma
Brief Title: Comparing 61.2 Gy Radiotherapy Dose Versus 50.4 Gy Radiotherapy Dose for Locally Advanced Esophageal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai 12
Record Dates: First submitted 2018-10-17; First posted 2018-12-31 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: chemoradiotherapy; esophageal cancer; PET/CT
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50.4Gy (Active Comparator): Total radiotherapy dose of 50.4Gy.
  Interventions: Radiation: Radiotherapy
- 61.2Gy (Experimental): Total radiotherapy dose of 61.2Gy.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Different total radiotherapy dose between two arms.

SUMMARY:
The purpose of this study is to determined the best definitive radiotherapy dosage for patients with locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75 years; both genders
* Esophageal squamous cell carcinoma confirmed by pathology.
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* Locally advanced esophageal squamous cell carcinoma (T1N1-3M0, T2-4NxM0, TxNxM1 (supraclavicular lymph node metastasis only) (AJCC 8th)
* Use of an effective contraceptive for adults to prevent pregnancy.
* No severely abnormal hematopoietic, cardiac, pulmonary, renal, or hepatic function. No immunodeficiency.
* WBC ≥ 3.5*109/L, Hemoglobin ≥ 9 g/dL, Neutrophils ≥ 1·5*109/L, Platelet count ≥ 100*109/L, ALAT and ASAT < 2·5 * ULN, TBIL < 1·5 * ULN, and Creatinine < 1·5 *ULN.
* ECOG 0-2.
* Life expectancy of more than 3 months.
* Agreement of PET/CT accessment at 25-28 radiotherapy fraction.

Exclusion Criteria:

* Total radiotherapy dose cannot reach 61.2Gy/34Fx in the condition of the nomal tissue dose complying to the standard criteria.
* Esophageal perforation, or hematemesis.
* History of radiotherapy or chemotherapy for esophageal cancer.
* History of surgery within 28 days before Day 1.
* History of prior malignancies (other than skin basal cell carcinoma or cervical carcinoma in situ with a disease-free survival of at least 3 years).
* Participation in other interventional clinical trials within 30 days.
* Pregnant or breast-feeding women or fertile patients who refused to use contraceptives.
* Drug addiction, alcoholism or AIDS.
* Uncontrolled seizures or psychiatric disorders.
* Any other condition which in the investigator's opinion would not make the patient a good candidate for the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival in PET/CT non-responders | 2 years
  The time between the start of the study treatment (Day 1) and death from any cause or last follow-up for patients alive at the end of the study.
Overall survival in ITT population | 2 years
  The time between the start of the study treatment (Day 1) and death from any cause or last follow-up for patients alive at the end of the study.

SECONDARY OUTCOMES:
Local control rate | 2 years
  The time between the start of the study treatment (Day 1) and local reccurence (included the primary tumor and regional lymph node failure)
Progression-free survival | 2 years
  (defined as the time between Day 1 and the first event of local failure, metastatic recurrence, progression or death)
Overall survival in PET/CT responders | 2 years
  Overall survival in patients who have SUV ≤ 4 in PET/CT analysis in 25-28 radiotherapy fractions.
Questionnaire EORTC-QLQ-C30 | 2 years
  A quality of life score is obtained according to the answers to the questionnaires.
Questionnaire EORTC-QLQ-OES18 | 2 years
  A quality of life score is obtained according to the answers to the questionnaires.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu H, Liu Q, Xu H, Mo M, Wang Z, Lu K, Zhou J, Chen J, Zheng X, Ye J, Ge X, Luo H, Liu Q, Deng J, Ai D, Hao S, Zhang J, Tseng IH, Song S, Chen Y, Zhao K. Dose escalation based on 18F-FDG PET/CT response in definitive chemoradiotherapy of locally advanced esophageal squamous cell carcinoma: a phase III, open-label, randomized, controlled trial (ESO-Shanghai 12). Radiat Oncol. 2022 Jul 29;17(1):134. doi: 10.1186/s13014-022-02099-y. PMID 35906623